CLINICAL TRIAL: NCT00002185
Title: A Pilot, Open-Label, Phase II, Randomized Study to Determine the Effects of Viracept on the Outcome of Cutaneous and Mucosal KS in AIDS Patients With CD4 <= 500 Cells/mm3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agouron Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 259F; AG1343-513
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-05

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Skin Neoplasms; AIDS-Related Opportunistic Infections; Sarcoma, Kaposi; Drug Therapy, Combination; HIV Protease Inhibitors; Mucous Membrane; Nelfinavir; Anti-HIV Agents
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Skin Neoplasms; AIDS-Related Opportunistic Infections | interventions — Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir mesylate

SUMMARY:
To determine the effect of Viracept in combination with modified antiretroviral therapy on the outcome of cutaneous and mucosal Kaposi's Sarcoma (KS).

DETAILED DESCRIPTION:
This is an open-label, randomized, pilot, Phase II study of the safety and efficacy of Viracept in combination with modified antiretroviral therapy as treatment in patients with cutaneous and mucosal KS. Patients will be randomized to modify (add or switch or initiate) their current antiretroviral therapy and will add Viracept or remain on their current background antiretroviral therapy for a 2 month period. Initially 20 patients will be randomized in a 2:1 ratio (i.e., 14 Viracept, 6 control) for a 2 month period. Response to therapy will be evaluated at the end of the 2 month control phase. At this point, patients who were initially assigned to the control arm will continue on open label Viracept for an additional 10 month period.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-positivity.
* Diagnosed KS proven by biopsy.
* NOTE:
* Patients must not opt for immediate topical, systemic or radiation treatment.
* At least 4 cutaneous lesions not treated within the previous 4 weeks.
* Life expectancy > 6 months.
* Signed, informed consent from parent or legal guardian for those patients < 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions and symptoms are excluded:

* Neoplastic disease (excluding KS) requiring systemic cytotoxic or radiation therapy or who have had these therapies within 1 month of baseline and have not completely recovered from the effects of these therapies.
* Unstable or severe intercurrent medical conditions, including but not limited to, significant symptomatic visceral KS.
* Clinically significant malabsorption syndrome.
* Renal insufficiency.

Patients with any of the following prior conditions are excluded:

Significant Fever (> 101 degrees F (38 degrees C) for >= 7 days) and/or diarrhea (> 6 loose stools/day for >= 7 days) within one month of baseline.

1. Immediate topical or systemic treatment for KS lesions.

* Use of Retinoid class drugs, either topically or systemically, or beta-carotene compounds or Vitamin A doses of more than 15,000 IU (5,000 mcg) per day concurrently.

Immediate radiation treatment.

1. Treatment of KS lesions with intra-lesional chemotherapy within 4 weeks of entry.

* History of > 2 weeks of prior therapy with Indinavir or Ritonavir.
* Use of Retinoid class drugs, either topically or systemically, or beta-carotene compounds or Vitamin A doses of more than 15,000 IU (5,000 mcg) per day within 4 weeks of entry.

Treatment of KS lesions with radiation within 4 weeks of entry. Active substance abusers; urine drug tests may be performed if drug abuse is suspected.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - LAC and USC Med Ctr / School of Medicine, Los Angeles, California
  - Univ of California / UCI Med Ctr, Orange, California
  - UCSD Treatment Ctr, San Diego, California
  - Santa Clara Valley Med Ctr, San Jose, California
  - Harbor - UCLA Med Ctr - Box 449, Torrance, California